CLINICAL TRIAL: NCT03157089
Title: LUX-Lung IO: A Phase II, Open Label, Non-randomised Study of Afatinib in Combination With Pembrolizumab in Patients With Locally Advanced or Metastatic Squamous Cell Carcinoma of the Lung
Brief Title: Testing Afatinib in Combination With Pembrolizumab in Patients With Squamous Cell Carcinoma of the Lung
Acronym: LUX-Lung-IO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1200-0283; 2016-005042-37 (EudraCT Number); PN497 (Other: Merck & Co.)
Record Dates: First submitted 2017-05-16; First posted 2017-05-17 (Actual); Results first posted 2021-02-23 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2021-02

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Afatinib; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- All patients (Experimental)
  Interventions: Drug: Afatinib; Drug: pembrolizumab

INTERVENTIONS:
Drug: Afatinib — Film-coated tablet
  Other Names: GILOTRIF, GIOTRIF, XOVOLTIB
Drug: pembrolizumab — Solution for infusion
  Other Names: KEYTRUDA®

SUMMARY:
The main objective is to assess the efficacy of afatinib in combination with pembrolizumab, as measured by objective response (OR) in patients with locally advanced or metastatic squamous NSCLC who progressed during or after first line platinum-based treatment.

The secondary objectives are to confirm the RP2D, assess the safety profile, and the secondary measures of clinical efficacy including disease control (DC), duration of objective response (DoR), progression-free survival (PFS), overall survival (OS), and tumour shrinkage.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed diagnosis of NSCLC considered to be of squamous histology, including mixed histology, in the opinion of the investigator.
* Locally advanced (stage IIIb) or metastatic (stage IV) NSCLC not considered eligible for curative therapy.
* Documented disease progression or relapse (based on investigator's assessment) during or after completion of at least 2 cycles of platinum-based chemotherapy as first line treatment of Stage IIIB/IV SCC of the lung. This includes patients relapsing within 6 months of completing (neo)adjuvant/curative-intent chemotherapy or definitive chemoradiotherapy. Patients should be eligible to receive 2nd line therapy in the opinion of the investigator.
* At least one target lesion (outside the brain) that can be accurately measured per Response Evaluation Criteria in Solid Tumours (RECIST) version 1.1. In patients who only have one target lesion and a biopsy of the lesion is required; the baseline imaging must be performed at least two weeks after the biopsy.
* Availability and willingness to provide a fresh tumour tissue sample obtained after relapse or progression on or after prior therapy. In case a fresh biopsy cannot be obtained (e.g. inaccessible lesions or patient safety concern), an archived specimen may be submitted.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Adequate organ function (all screening labs should be performed within 10 days prior to treatment initiation).
* Recovery from major surgery or any previous anti-cancer or radiation therapy-related toxicity to ≤ CTCAE Grade 1 at C1_V1 (except for alopecia; stable sensory neuropathy must be ≤ CTCAE Grade 2).
* At least 18 years of age or over the legal age of consent in countries where that is greater than 18 years at screening.
* Signed and dated written informed consent in accordance with ICH-GCP and local legislation prior to admission to the trial.
* Male or female patients. Women of childbearing potential (WOCBP) and men able to father a child must be ready and able to use highly effective methods of birth control per ICH M3 (R2) that result in a low failure rate of less than 1% per year when used consistently and correctly, starting with the screening visit and through 120 days after the last dose of pembrolizumab treatment and 2 weeks after last afatinib treatment, respectively, as listed in the protocol. A list of contraception methods meeting these criteria is provided in the patient information.

  * Note: Female patients of childbearing potential must have a negative urine or serum pregnancy test within 72 hours prior to taking study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required. The serum pregnancy test must be negative for the patient to be eligible.

Exclusion criteria:

* Prior therapy with any immune checkpoint inhibitor; however, prior (neo) adjuvant checkpoint inhibitor therapy is allowed if completed at least 12 months before relapse.
* Prior therapy with EGFR inhibiting drugs; however, prior EGFR-targeted (neo) adjuvant therapy is allowed if completed at least 12 months before relapse.
* Treatment with prior chemotherapy, non-EGFR targeted therapy, or anti-cancer hormonal treatment within 2 weeks prior to the first dose of trial treatment.
* Current or previous treatment with experimental therapy or use of an investigational device within 30 days prior to the first dose of trial treatment.
* Prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to the first dose of trial treatment.
* Received a live vaccine within 30 days prior to the first dose of trial treatment. Seasonal flu vaccines that do not contain live virus are permitted.
* Diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment. The use of physiologic doses of corticosteroids is allowed.
* Any history of or concomitant condition that, in the opinion of the investigator, would compromise the patient's ability to comply with the trial or interfere with the evaluation of the efficacy and safety of the test drugs.
* Radiotherapy within 4 weeks prior to start of treatment except as follows:

  * Palliative radiotherapy to regions other than the chest is allowed up to 2 weeks prior to start of treatment;
  * Single dose palliative radiotherapy for symptomatic metastasis within 2 weeks prior to start of treatment may be allowed but must be agreed with the Sponsor.
* Major surgery (according to the investigator's assessment) performed within 4 weeks prior to start of treatment or planned during the projected course of the study.
* Requirement or wish to continue the intake of restricted medications or any drug considered likely to interfere with the safe conduct of the trial.
* Known history of hypersensitivity to afatinib or any of its excipients.
* Known history of hypersensitivity (≥Grade 3) to pembrolizumab and/or any of its excipients.
* Known active central nervous system (CNS) metastases and/or carcinomatous meningitis.

  -- Note: Patients with previously treated brain metastases may participate provided they are radiologically stable i.e. without evidence of progression for at least four weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable, and without requirement of steroids treatment for at least 14 days prior to first dose of study treatment. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability.
* Active autoimmune disease that has required systemic treatment in past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g. thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment and is allowed.
* History of (non-infectious) interstitial lung disease (ILD)/pneumonitis that required steroids or current ILD/pneumonitis.
* Any history or presence of uncontrolled gastrointestinal disorders that could affect the intake and/or absorption of the study drug (e.g. nausea, vomiting, Crohn's disease, ulcerative colitis, chronic diarrhoea, malabsorption) in the opinion of the investigator.
* Active infectious disease requiring systemic therapy or which puts the patient at increased risk in the opinion of the investigator.
* Previous or concomitant malignancies at other sites than the lung, except:

  * Effectively treated non-melanoma skin cancers;
  * Effectively treated carcinoma in situ of the cervix;
  * Effectively treated ductal carcinoma in situ;
  * Other effectively treated malignancy that has been in remission for more than 3 years and is considered to be cured.
* Known human immunodeficiency virus (HIV) (HIV 1/2 antibodies), hepatitis B (e.g. HBsAg reactive) or known active hepatitis C infection.
* History of active TB (Bacillus Tuberculosis).
* History or presence of cardiovascular abnormalities such as uncontrolled hypertension, congestive heart failure New York Heart Association (NYHA) classification of ≥3, unstable angina or poorly controlled arrhythmia which are considered as clinically relevant by the investigator. Myocardial infarction within 6 months prior to start of treatment.
* Psychiatric, substance abuse disorders, or chronic alcohol abuse or any condition as per investigator's opinion.
* Further criteria apply, some were shortened.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-11-02 (Actual); Primary Completion 2020-01-13 (Actual); Study Completion 2020-01-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (13):
- Baptist Health Medical Group, Lexington, Kentucky, United States
- France (4):
  - HOP Côte de Nacre, Caen
  - HOP Le Mans, Le Mans
  - HOP Nord, Marseille
  - HOP Nord Laënnec, Nantes
- South Korea (2):
  - Severance Hospital, Seoul
  - Asan Medical Center, Seoul
- Spain (4):
  - Hospital Vall d'Hebron, Barcelona
  - Complejo Hospitalario Universitario Insular - Materno Infantil, Las Palmas de Gran Canaria
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Clínico Universitario Lozano Blesa, Zaragoza
- Turkey (Türkiye) (2):
  - Hacettepe Universitesi Tip Fakultesi, Onkoloji ABD, Ankara
  - Istanbul Universitesi Cerrahpasa Tip Fakultesi, Istanbul

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Levy B, Barlesi F, Paz-Ares L, Bennouna J, Erman M, Felip E, Isla D, Ryun Kim H, Kim SW, Madelaine J, Molinier O, Ozguroglu M, Rodriguez Abreu D, Adeniji A, Lorence RM, Voccia I, Chisamore MJ, Riess JW. Phase II study of afatinib plus pembrolizumab in patients with squamous cell carcinoma of the lung following progression during or after first-line chemotherapy (LUX-Lung-IO). Lung Cancer. 2022 Apr;166:107-113. doi: 10.1016/j.lungcan.2022.01.023. Epub 2022 Feb 3. PMID 35257949
- [Derived] Levy B, Paz-Ares L, Bennouna J, Felip E, Abreu DR, Isla D, Barlesi F, Molinier O, Madelaine J, Audigier-Valette C, Kim SW, Kim HR, Ozguroglu M, Erman M, Badin FB, Mekhail TM, Scheff R, Chisamore MJ, Sadrolhefazi B, Riess JW. Afatinib With Pembrolizumab for Treatment of Patients With Locally Advanced/Metastatic Squamous Cell Carcinoma of the Lung: The LUX-Lung IO/KEYNOTE 497 Study Protocol. Clin Lung Cancer. 2019 May;20(3):e407-e412. doi: 10.1016/j.cllc.2018.12.022. Epub 2019 Jan 4. PMID 30808583
- See also: Related Info — http://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This trial is an open-label, single arm phase II study assessing the tolerability and anti-tumour activity of afatinib when given in combination with a fixed dose of pembrolizumab in patients with locally advanced or metastatic squamous non-small-cell lung cancer (NSCLC), who progressed during or after first line platinum-based standard therapy and had no prior treatment with an immune checkpoint inhibitor or Epidermal Growth Factor Receptor (EGFR) targeted therapy.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria. Subjects were not to be allocated to a treatment group, if any of the entry criteria were violated.
  The trial consisted of 2 parts: A safety run-in and the main part. After the safety run-in, a safety-monitoring committee (SMC) decided not to proceed with the main part.
Groups:
- Afatinib 40 mg + Pembrolizumab 200 mg: 40 milligram (mg) of afatinib film-coated tablet, given orally with a glass of water (without food consumption 3 hours (h) prior and 1h post afatinib administration), once daily + pembrolizumab 200 mg, intravenous infusion, once every 3 weeks.
  Both afatinib and pembrolizumab were to be given until documented disease progression, or unacceptable adverse events, or other reasons requiring treatment discontinuation, or for up to 35 cycles of 21 days (i.e. the approved pembrolizumab monotherapy duration). In case of early discontinuation of one agent, the other agent could be continued as monotherapy for altogether up to 35 cycles.
- Afatinib 30 mg + Pembrolizumab 200 mg: 30 mg of afatinib film-coated tablet, given orally with a glass of water (without food consumption 3 hours (h) prior and 1h post afatinib administration), once daily + pembrolizumab 200 mg, intravenous infusion, once every 3 weeks.
  Both afatinib and pembrolizumab were to be given until documented disease progression, or unacceptable adverse events, or other reasons requiring treatment discontinuation, or for up to 35 cycles of 21 days (i.e. the approved pembrolizumab monotherapy duration). In case of early discontinuation of one agent, the other agent could be continued as monotherapy for altogether up to 35 cycles.
Period: Overall Study
Arm/Group | Afatinib 40 mg + Pembrolizumab 200 mg | Afatinib 30 mg + Pembrolizumab 200 mg
Started | 12 | 12
Treated (Treated with afatinib+pembrolizumab) | 12 | 12
Completed | 0 | 0
Not Completed | 12 | 12
Not completed — Treated only with pembrolizumab | 1 | 0
Not completed — Adverse Event | 5 | 4
Not completed — Progressive disease | 6 | 8

BASELINE CHARACTERISTICS:
Population: The treated set (TS) included all participants, who received at least one dose of afatinib or pembrolizumab.
Groups:
- Total: Total of all reporting groups
Arm/Group | Afatinib 40 mg + Pembrolizumab 200 mg | Afatinib 30 mg + Pembrolizumab 200 mg | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.8 (10.0) | 63.3 (7.3) | 63.1 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 5
  Male | 8 | 11 | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 5 | 0 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 6 | 8 | 14
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 4 | 5

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: Objective response rate is defined as percentage of participants with the best overall response of complete response (CR, disappearance of all target lesions) or confirmed partial response (PR, at least a 30% decrease in sum of diameter (SoD, longest diameter (LD) measured for all lesions except lymph nodes, where shortest diameter (ShD) was used) of target lesions, reference is baseline SoD). Tumour response was assessed based on local radiological image (Computerised tomography (CT) or Magnetic resonance imaging (MRI)) evaluation by the investigators according to Response Evaluation Criteria In Solid Tumours (RECIST) version 1.1.
Time Frame: Tumour assessment performed at screening (-28 days), week 9 (day 56-63) after study treatment (afatinib or pembrolizumab) start and every 9th week thereafter, up to 556 days.
Population: The treated set (TS) included all participants, who received at least one dose of afatinib or pembrolizumab.
Measure: Number; unit: Percentage of Participants
Arm/Group | Afatinib 40 mg + Pembrolizumab 200 mg | Afatinib 30 mg + Pembrolizumab 200 mg
Number analyzed (Participants) | 12 | 12
Percentage of Participants | 16.7 | 8.3

2. Secondary Outcome: Recommended Phase II Dose (RP2D)
Description: Recommended Phase II Dose (RP2D) was to be calculated through a Bayesian logistic regression model (BLRM) with overdose control that was to be fitted to binary toxicity outcomes. After 12 patients had completed at least one cycle (one cycle equals 21 days and consists of one time infusion of pembrolizumab at Day 1 + daily intake of afatinib) of treatment, the prior distributions were to be updated through Gibbs sampling procedures with the accumulated dose limiting toxicity (DLT) data from the first treatment cycle. The estimate of parameters was to be updated as data were accumulated using the BLRM. At the end of the dose confirmation, the toxicity probability at each dose level was to be calculated to determine an estimate of the RP2D. Posterior probabilities for the rate of DLT were to be summarised from BLRM. Confirmation of the RP2D by the Safety Monitoring Committee (SMC) was to be based on these probabilities as well as on the review of other safety and laboratory data.
Time Frame: 21 days (1 treatment cycle) from study treatment (afatinib and pembrolizumab) administration.
Population: The treated set (TS) included all participants, who received at least one dose of afatinib or pembrolizumab. Because the Safety Monitoring Committee (SMC) decided that the benefit-risk ratio of afatinib in combination with pembrolizumab was not favorable, the trial was stopped according to a protocol-defined option and the decision on RP2D was not performed.
Measure: Number; unit: Milligramm (mg)
Groups:
- Afatinib + Pembrolizumab: Comprises both arms during the safety run-in part. 30 or 40 milligram (mg) of afatinib film-coated tablet, given orally with a glass of water (without food consumption 3 hours (h) prior and 1h post afatinib administration), once daily + pembrolizumab 200 mg, intravenous infusion, once every 3 weeks.
  Both afatinib and pembrolizumab were to be given until documented disease progression, or unacceptable adverse events, or other reasons requiring treatment discontinuation, or for up to 35 cycles of 21 days (i.e. the approved pembrolizumab monotherapy duration). In case of early discontinuation of one agent, the other agent could be continued as monotherapy for altogether up to 35 cycles.
Arm/Group | Afatinib + Pembrolizumab
Number analyzed (Participants) | 24
Milligramm (mg) | NA — Because the Safety Monitoring Committee (SMC) decided that the benefit-risk ratio of afatinib in combination with pembrolizumab was not favorable, the trial was ended according to a protocol-defined option and the decision on RP2D was not performed.

3. Secondary Outcome: Disease Control Rate (DCR)
Description: Disease control rate was calculated as percentage of participants with CR, PR, or stable disease (SD, neither sufficient shrinkage to qualify for PR, taking as reference the baseline sum of diameters (SoD), nor sufficient increase to qualify for progressive disease (PD, at least a 20% increase in the SoD of target lesions, taking as reference the smallest SoD recorded on study (including baseline), together with an absolute increase in the SoD of at least 5 millimeter (mm ) or the appearance of one or more new lesions). Tumour response was assessed based on local radiological image (Computerised tomography (CT) or Magnetic resonance imaging (MRI)) evaluation by the investigators according to Response Evaluation Criteria In Solid Tumours (RECIST) version 1.1.
Time Frame: as for outcome 1
Population: The treated set (TS) included all participants who received at least one dose of afatinib or pembrolizumab.
Measure: Number; unit: Percentage of participants
Arm/Group | Afatinib 40 mg + Pembrolizumab 200 mg | Afatinib 30 mg + Pembrolizumab 200 mg
Number analyzed (Participants) | 12 | 12
Percentage of participants | 50 | 58.3

4. Secondary Outcome: Duration of Objective Response (DOR)
Description: For participants who showed objective response, duration of objective response (DoR), was defined as the time from first documented complete response (CR) or partial response (PR) until the earliest of disease progression (PD) or death. Tumour response was assessed based on local radiological image (CT or MRI) evaluation by the investigators according to RECIST version 1.1. The number of participants with objective response who experienced the event "disease progression or death (whichever came first)" is reported instead of a metric summarizing the time-to-event data with unit of time, as the number analyzed was too small to perform a Kaplan-Meier-analysis.
Time Frame: Tumour assessment performed at screening (-28 days), week 9 (day 56-63) after study treatment (afatinib or pembrolizumab) start and every 9th week thereafter, up to 436 days.
Population: All participants who received at least one dose of afatinib or pembrolizumab and showed objective response.
Measure: Count of Participants; unit: Participants
Arm/Group | Afatinib 40 mg + Pembrolizumab 200 mg | Afatinib 30 mg + Pembrolizumab 200 mg
Number analyzed (Participants) | 2 | 1
Participants | 2 | 1

5. Secondary Outcome: Progression-free Survival (PFS)
Description: Progression-free survival was defined as the time (weeks) from the date of the first afatinib or pembrolizumab administration to the date of disease progression (at least a 20% increase in the sum of diameter (SoD, longest diameter (LD) measured for all lesions except lymph nodes, where shortest diameter (ShD) was used) of target lesions, taking as reference the smallest SoD recorded on study (including baseline), together with an absolute increase in the SoD of at least 5 mm or the appearance of one or more new lesions) or death (if the patient died without progression). The date of progression for the primary analyses was determined based on investigator assessment. Tumour response was assessed based on local radiological image (Computerised tomography (CT) or Magnetic resonance imaging (MRI)) evaluation by the investigators according to RECIST version 1.1. Median and 95% Confidence Interval were calculated using Kaplan-Meier estimates.
Time Frame: as for outcome 1
Population: The treated set (TS) included all participants, who received at least one dose of afatinib or pembrolizumab.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Afatinib 40 mg + Pembrolizumab 200 mg | Afatinib 30 mg + Pembrolizumab 200 mg
Number analyzed (Participants) | 12 | 12
weeks | 9.0 [4.6 to 27.1] | 14.4 [5.0 to 26.1]

6. Secondary Outcome: Overall Survival (OS)
Description: Overall survival is defined as the time from the date of treatment start to the date of death from any cause. Participants without event were censored. Median and 95% Confidence Interval were calculated using Kaplan-Meier estimates.
Time Frame: From Day 1 of study treatment (afatinib or pembrolizumab) administration up to a total of 574 days.
Population: The treated set (TS) included all participants, who received at least one dose of afatinib or pembrolizumab.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Afatinib 40 mg + Pembrolizumab 200 mg | Afatinib 30 mg + Pembrolizumab 200 mg
Number analyzed (Participants) | 12 | 12
weeks | 37.9 [15.0 to 59.3] | 26.6 [8.6 to 53.6]

7. Secondary Outcome: Tumour Shrinkage
Description: Tumour shrinkage (in millimeters) is defined as the difference between the minimum post-baseline sum of diameters of target lesions (SoD, longest for non-nodal lesions, short axis for nodal lesions) and the baseline sum of diameters of the same set of target lesions. Tumour shrinkage is reported as percentage change from baseline and represents the maximum decrease or the minimum increase from baseline in SoD in percentage of the baseline SoD. Negative values indicate a reduction in the SoD; positive values indicate an increase in the SoD. Tumour response was assessed based on local radiological image (CT or MRI) evaluation by the investigators according to RECIST 1.1.
Time Frame: as for outcome 1
Population: The treated set (TS) included all participants, who received at least one dose of afatinib or pembrolizumab.
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Afatinib 40 mg + Pembrolizumab 200 mg | Afatinib 30 mg + Pembrolizumab 200 mg
Number analyzed (Participants) | 12 | 12
Percentage change | -7.7 (29.83) | 22.0 (71.84)

ADVERSE EVENTS:
Time Frame: [Timeframe for All-Cause Mortality]: From Day 1 of study treatment (afatinib or pembrolizumab) administration up to a total of 574 days. [Timeframe for Serious and Other Adverse Events]: From the time of first drug administration till the end of treatment + 30 days residual effect period (REP), up to 558 days.
Description: The treated set (TS) included all participants, who received at least one dose of afatinib or pembrolizumab.
Arm/Group | Afatinib 40 mg + Pembrolizumab 200 mg | Afatinib 30 mg + Pembrolizumab 200 mg
All-Cause Mortality (participants affected / at risk) | 10/12 | 10/12
Serious Adverse Events (participants affected / at risk) | 4/12 | 9/12
Other Adverse Events (participants affected / at risk) | 12/12 | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Afatinib 40 mg + Pembrolizumab 200 mg (N=12) | Afatinib 30 mg + Pembrolizumab 200 mg (N=12)
Acute coronary syndrome (Cardiac disorders) | 0 | 1
Pericardial effusion (Cardiac disorders) | 1 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1
Multiple organ dysfunction syndrome (General disorders) | 1 | 0
Immune-mediated hepatitis (Hepatobiliary disorders) | 0 | 1
Bronchitis (Infections and infestations) | 0 | 3
Pneumonia (Infections and infestations) | 1 | 1
Blood bilirubin increased (Investigations) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Immune-mediated pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Extremity necrosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Afatinib 40 mg + Pembrolizumab 200 mg (N=12) | Afatinib 30 mg + Pembrolizumab 200 mg (N=12)
Anaemia (Blood and lymphatic system disorders) | 3 | 3
Atrial fibrillation (Cardiac disorders) | 1 | 0
Hyperthyroidism (Endocrine disorders) | 2 | 2
Hypothyroidism (Endocrine disorders) | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Cheilitis (Gastrointestinal disorders) | 2 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 11 | 7
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 4
Stomatitis (Gastrointestinal disorders) | 4 | 1
Vomiting (Gastrointestinal disorders) | 3 | 3
Asthenia (General disorders) | 2 | 3
Chest pain (General disorders) | 1 | 1
Face oedema (General disorders) | 0 | 1
Fatigue (General disorders) | 3 | 4
Mucosal inflammation (General disorders) | 1 | 2
Non-cardiac chest pain (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 1 | 1
Pyrexia (General disorders) | 2 | 0
Vessel puncture site swelling (General disorders) | 1 | 0
Cholestasis (Hepatobiliary disorders) | 1 | 0
Hepatic pain (Hepatobiliary disorders) | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1
Hepatitis viral (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 0
Paronychia (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 1
Subcutaneous abscess (Infections and infestations) | 0 | 1
Tracheobronchitis (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 1
Amylase increased (Investigations) | 3 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 2 | 0
Blood creatinine increased (Investigations) | 1 | 2
Gamma-glutamyltransferase increased (Investigations) | 2 | 1
International normalised ratio increased (Investigations) | 1 | 0
Lipase increased (Investigations) | 1 | 1
Lymphocyte count decreased (Investigations) | 1 | 0
Transaminases increased (Investigations) | 1 | 0
Weight decreased (Investigations) | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 6 | 3
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 2
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Tendon pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Dysgeusia (Nervous system disorders) | 0 | 1
Neuralgia (Nervous system disorders) | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 1
Depression (Psychiatric disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 1
Pelvic pain (Reproductive system and breast disorders) | 0 | 1
Prostatitis (Reproductive system and breast disorders) | 0 | 1
Aphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Restrictive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 1 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 2 | 5
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 1
Rash (Skin and subcutaneous tissue disorders) | 5 | 1
Skin erosion (Skin and subcutaneous tissue disorders) | 1 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 1
Xeroderma (Skin and subcutaneous tissue disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
After the safety run-in, the SMC decided that the benefit-risk ratio was not favorable and recommended ending the trial according to a protocol-defined option. Trial was completed as described in protocol.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-05-14): https://cdn.clinicaltrials.gov/large-docs/89/NCT03157089/SAP_000.pdf
  • Study Protocol (2019-04-11): https://cdn.clinicaltrials.gov/large-docs/89/NCT03157089/Prot_002.pdf